CLINICAL TRIAL: NCT05031884
Title: Vision-based Ultrasonic Robot Autonomous Scanning Research
Status: Not yet recruiting | Type: Observational
Sponsor: Rongqin Zheng (Other)
Responsible Party: Sponsor-Investigator, Rongqin Zheng, Professors, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: sysu-robot 2021
Record Dates: First submitted 2021-08-29; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Ultrasound Therapy; Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MGIR3-US group: using MGIR3-US to do ultrasonic examinations.
  Interventions: Device: MGIR3-US
- control group: using conventional B-mode ultrasound to do ultrasonic examinations.

INTERVENTIONS:
Device: MGIR3-US — MGIR3-US is an remote scanning robot which can do ultrasonic examinations.
  Groups: MGIR3-US group

SUMMARY:
MGIR3-US is a remote scanning robot which can perform ultrasound exam. The aim of the study is to evaluate the feasibility and the application of MGIR3-US.

ELIGIBILITY:
Inclusion Criteria:

* patients who agree using MGIR3 to do ultrasonic examinations
* age from 18 to 65

Exclusion Criteria:

* Patients who has trauma on the inspection site or on the body surface
* Pregnant patients.
* Patients who are afraid of MGIR3-US

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers are encouraged in the study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-08-31 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The degree of satisfaction in participants | from 2021.08 to 2024.08
  The degree of satisfaction in participants

SECONDARY OUTCOMES:
The degree of satisfaction in doctors | from 2021.08 to 2024.08
  The degree of satisfaction in doctors
the lesion inspection rate | from 2021.08 to 2024.08
  the lesion inspection rate

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ren, doctor, Principal Investigator — the third affiated hosptial of Sun Yat-sun University
Locations (1):
- Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided